CLINICAL TRIAL: NCT04163770
Title: Evaluation Of Performance & Complications of Pacemakers in Children
Brief Title: Evaluation Of Pacemakers in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, khaled mohammed allam, assistant lecturer of pediatric, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: EPCP
Record Dates: First submitted 2019-10-28; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Disorder of Cardiac Pacemaker System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- performance of pacemaker at time of implantation (Experimental)
  Interventions: Device: caliberation of pacemaker
- performance of pacemaker 6 months after implantation (Experimental)
  Interventions: Device: caliberation of pacemaker

INTERVENTIONS:
Device: caliberation of pacemaker — evaluation of ventricular impedence, ventricular sensing, ventricular capture threshold
  Arms: performance of pacemaker at time of implantation
Device: caliberation of pacemaker — evaluation of ventricular impedence, ventricular sensing, ventricular capture threshold
  Arms: performance of pacemaker 6 months after implantation

SUMMARY:
Pacemakers were introduced into clinical practice several decades ago and currently are used in a growing number of patients. Since insertion of the first cardiac Pacemaker in 1958, vast changes have occurred in both the technology of the devices and their indications. Devices have evolved from single-lead and fixed-rate systems to multi chamber rate-responsive systems with increasingly sophisticated software .

Pediatric Pacemaker implants comprise less than 1 % of all implants. The indications for pacing in newborns and infants are divided predominantly into three groups: congenital abnormalities of the conduction system, acquired heart blocks after cardiac surgery for correction of congenital defects, and sinus node diseases

DETAILED DESCRIPTION:
Although advances in device and lead technology have expanded the ability to implant pacemakers and defibrillators in children and patients with congenital heart disease , a number of challenges exist that can complicate long-term pacing success in this unique population . These include a long duration of pacing need, a more active lifestyle in young patients, somatic growth, congenital cardiac abnormalities, and relatively small patient and vessel size. Traditional stylet driven leads have limited maneuverability, making lead placement in smaller patients and those with structural abnormalities more challenging.

Additionally, the larger lead diameter needed to accommodate the stylet has been correlated with increased risk of venous complications in children . Furthermore, many congenital heart disease patients have structural abnormalities and cardiac scarring that require pacing leads to be placed in non-standard locations, and selective site pacing can be difficult to achieve with stylet-driven leads .

Pacing therapy in children must take into account several unique pediatric issues: (1) small physique; (2) somatic growth; (3) presence of intracardiac shunts; and (4) a complex anatomical heart structure. It is important to understand these features when deciding whether pacing is indicated, as well as when selecting the time to implant and how to implant.

The 2008 Guidelines of the American College of Cardiology /American Heart Association /Heart Rhythm Society summarize indications for pacing treatment in children. Atrioventricular block including congenital atrioventricular block associated with cardiac surgery or a natural history of complex congenital heart disease such as corrected transposition of the great arteries are the most important indications for pacemaker implantation in children 8-13. In pediatric patients, atrioventricular block that does not recover within 7-10 days after cardiac surgery is associated with a risk of sudden cardiac death in the future, so pacemaker implantation is recommended.

Dual-chamber pacemakers are often selected for adult patients with atrioventricular block. Dual-chamber pacemakers pacing requires two endocardial leads. In infants, this presents a problem because the venous diameter is small and may cause venous obstruction. A single chamber ventricular pacemaker instead of a dual-chamber pacemaker is a good alternative choice in children with complete atrioventricular block and normal sinus node function, because it requires only a single lead and may reduce the possibility of venous occlusion. The high heart rate of infants is another issue. The mean heart rate of an infant is 100 bpm or faster, increasing to 180-200 bpm or above when crying. In an infant with atrioventricular block, the atrial rate becomes so rapid that it may exceed the maximum programmable upper tracking rate, which is limited by the post-ventricular atrial refractory period and atrioventricular delay. Under the condition where the atrial heart rate exceeds the maximum programmable upper tracking rate, symptomatic 2:1 atrioventricular block may occur. Therefore, in infants with a small body size and a rapid ventricular rate, single chamber ventricular pacing or single-chamber ventricular pacing with rate response should be selected.

ELIGIBILITY:
Inclusion Criteria:

• Pediatric age group 0 month -18 years Indicated for permanent cardiac pacing

Exclusion Criteria:

* Cardiomyopathy unrelated to rhythm disturbance.
* Significant systemic disease apart from the cardiac one

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-15 (Estimated); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
Performance of pacemakers in children | 1 year
  the performance will be assessed by Ventricular impedence in ohms
Performance of pacemakers in children | 1 year
  the performance will be assessed by ventricular capture threshold in volt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garnreiter J, Whitaker P, Pilcher T, Etheridge S, Saarel E. Lumenless pacing leads: performance and extraction in pediatrics and congenital heart disease. Pacing Clin Electrophysiol. 2015 Jan;38(1):42-7. doi: 10.1111/pace.12508. Epub 2014 Sep 16. PMID 25224253